CLINICAL TRIAL: NCT01870531
Title: Transient Ischemic Attacks in Korean: Hospital-based, Multi-center Prospective Registry
Brief Title: Korean Transient Ischemic Attack eXpression Registry
Acronym: KTX registry
Status: Completed | Type: Observational
Sponsor: Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, Yong-Seok Lee, Professor, Seoul National University Boramae Hospital
Other Study IDs: 800-20100046
Record Dates: First submitted 2013-05-23; First posted 2013-06-06 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Transient Ischemic Attack
Keywords: Transient Ischemic Attack
MeSH Terms: conditions — Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to determine the clinical and neuroimaging characteristics of Transient Ischemic Attacks in Korean populations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms and signs consistent with transient ischemic attack
* Subject who admitted hospital within 24 hours after symptom onset
* Subjects who underwent MRI (including diffusion-weighted images) and MRA (or CT angiography)

Exclusion Criteria:

Transient neurological symptoms due to

* Migraine aura
* Basilar migraine
* Seizures
* Syncope
* Peripheral vertigo
* Transient global amnesia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University Hospitals
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Vascular events including ischemic strokes, myocardial infarctions, cardiovascular deaths | 90 days

SECONDARY OUTCOMES:
Recurrent transient ischemic attacks | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Seok Lee, MD, PhD, Principal Investigator — Seoul National University Boramae Hospital
Locations (1):
- Seoul National University Boramae Hospital, Seoul, Seoul, South Korea